CLINICAL TRIAL: NCT02150447
Title: Effect of Proton Pump Inhibitor on Prevention of Tumor Bleeding in Patients Under Palliative Chemotherapy for Unresectable Gastric Cancer: a Randomized, Double Blind, and Placebo Controlled Multicenter Trial
Brief Title: The Use of Proton Pump Inhibitor on the Prevention of Gastric Cancer Bleeding
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enroll rate
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Pusan National University Hospital (Other); Kosin University Gospel Hospital (Other); Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, Il Ju Choi, Head of Gastric Cancer Cencer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCCCTS09420; 0910090 (Other Grant/Funding Number: National Cancer Center, Korea); 1210520 (Other Grant/Funding Number: National Cancer Center, Korea)
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Gastric Cancer; Bleeding
Keywords: Gastric cancer bleeding; Proton pump inhibitor
MeSH Terms: conditions — Stomach Neoplasms; Hemorrhage | interventions — Proton Pump Inhibitors; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator): Proton pump inhibitor (lansoprazole) therapy for the prevention of gastric cancer bleeding
  Interventions: Drug: Proton pump inhibitor
- Placebo group (Placebo Comparator): Placebo for the prevention of gastric cancer bleeding
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proton pump inhibitor — Lansoprazole 30 mg, daily
  Other Names: Lansoprazole
  Arms: Intervention group
Drug: Placebo — Placebo, daily
  Arms: Placebo group

SUMMARY:
The aim of this study is the effect of proton pump inhibitor (PPI) with respect to gastric cancer bleeding in inoperable patients.

DETAILED DESCRIPTION:
Tumor bleeding frequently occurs in inoperable gastric cancer patients. Inoperable gastric cancer usually has a large ulcer with friable tumor vessels. Acidic environment in stomach prevents adequate function of coagulation cascade and decrease clot stability. Gastric cancer bleeding may cause significant morbidity and often delays scheduled chemotherapy. National Center Center data showed that about 30% of gastric cancer patient undergoing palliative chemotherapy eventually experience significant cancer bleeding during the treatment period. Once bleeding occurs, endoscopic management is more difficult in gastric cancer patients than in patients with benign peptic ulcers, because the malignant ulcer bed has significant fibrosis. Consequently, gastric cancer patient has a high risk of rebleeding.

Proton pump inhibitor (PPI, lansoprazole for example) decrease gastric acid secretion by inhibiting H+,K+-ATPase, and subsequently stabilize blood clot. PPIs are commonly used for benign peptic ulcer or reflux esophagitis, and PPI can decrease recurrent benign ulcer bleeding or other ulcer complications. Moreover, it was reported to prevent bleeding from NSAID or aspirin induced gastric ulcer. Because PPIs are very safe, and they are even available as over-the-counter drugs in some countries. Furthermore, the drug has no interaction with major chemotherapeutic agents commonly used for gastric cancer. Moreover, the drugs are prescribed to the gastric cancer patients when tumor bleeding occurs. Although gastric cancer bleeding is not uncommon and clinically challenging problem, there has been no recommended measure to prevent cancer bleeding. Also there has been no report about the efficacy of PPIs on the gastric cancer bleeding prevention up to now.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary gastric adenocarcinoma
* Age ≥18 years
* Plan for 1st line or 2nd line palliative chemotherapy
* Cancer staging: metastatic (TxNxM1) or locally advanced unresectable gastric cancer (T4NxMx with unresectable), or T2-3NxMx with inoperable condition
* Performance status (PS) of 0 to 2 on Eastern Cooperative Oncology Group (ECOG) scale
* Adequate organ functions defined as indicated below: (a) WBC > 3000/mm3, (b) Hb 9.0 g/dL regardless of any transfusion history, (c) Platelet ≥100,000/mm3, (d) AST/ALT ≤ 2.5 x UNL (≤ 5 x UNL if liver metastases are present) (e) Total bilirubin ≤1.5x UNL (f) Cr ≤1.5 x UNL
* Written informed consent

Exclusion Criteria:

* Other malignancy within the past 3 years except adequately treated non-melanomatous skin cancer or carcinoma in situ of the cervix
* Patients with significant or uncontrolled gastrointestinal bleeding in the past two weeks without evidence of resolution documented by endoscopy or colonoscopy
* Previous subtotal gastrectomy or total gastrectomy
* Patient with a plan for neo-adjuvant chemotherapy
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome, or inability to take oral medication
* Allergy history to proton pump inhibitor
* Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
* Inadequate cardiovascular function: (a) New York Heart Association class III or IV heart disease, (b) Unstable angina or myocardial infarction within the past 6 months, (c) History of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality
* Requirement for therapeutic anticoagulant therapy, aspirin or non-steroidal anti-inflammatory agents except COX-2 selective inhibitor
* Requirement for therapeutic corticosteroid; the use of dexamethasone as anti-emetics or a premedication of chemotherapy-associated hypersensitivity is not an exclusion criteria
* Need for PPI maintenance treatment for uncontrolled reflux esophagitis or active peptic ulcer
* Psychiatric disorder that would preclude compliance
* Pregnant or breast-feeding women
* Untreated folate or vitamine B12 deficiency anemia
* Bone marrow metastasis, or evidence of microangiopathic hemolytic anemia (MAHA)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2009-06; Primary Completion 2015-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Time-to-bleeding event | Up to 6 years of study period
  Evaluation of the effect of PPI on the prevention of gastric cancer bleeding

SECONDARY OUTCOMES:
Transfusion requirement (packed RBC unit) | Up to 6 years of study period
  Unit of packed RBC required at the time of tumor bleeding
Number of endoscopy to evaluate tumor bleeding | Up to 6 years of study period
  No of endoscopic session to evaluation bleeding from advanced gastric cancer
Number of endoscopic treatment for cancer bleeding | Up to 6 years of study period
  Total number of endoscopic treatment perfomed for gastric cancer bleeding in each patient
Overall survival | Up to 6 years of study period

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, M.D., Ph.D., Principal Investigator — National Cancer Center, Korea; Gwang Ha Kim, M.D., Ph.D., Principal Investigator — Pusan National University Hospital; Moo In Park, M.D., Ph.D., Principal Investigator — Kosin University Gospel Hospital; Won Sup Lee, M.D., Ph.D., Principal Investigator — Gyeongsang National University Hospital
Locations (4):
- South Korea (4):
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang
  - Gyeong Sang National University Hospital, Jinju

REFERENCES:
- [Derived] Kim YI, Kim MJ, Park SR, Kim HK, Cho SJ, Lee JY, Kim CG, Kim GH, Park MI, Nam BH, Park YI, Choi IJ. Effect of a Proton Pump Inhibitor on Tumor Bleeding Prevention in Unresectable Gastric Cancer Patients: a Double-Blind, Randomized, Placebo-Controlled Trial. J Gastric Cancer. 2017 Jun;17(2):120-131. doi: 10.5230/jgc.2017.17.e15. Epub 2017 May 31. PMID 28680717